CLINICAL TRIAL: NCT07011199
Title: Evaluation of Clinical Outcomes in Biliary Atresia Patients Undergoing Kasai Surgery Before 90 Days of Age With Umbilical Cord-Derived Mesenchymal Stem Cell Therapy
Brief Title: Clinical Outcomes of Early Kasai Surgery With Umbilical Cord MSCs in Biliary Atresia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Avriana Pety Wardani, MD, Sp. BA, Dr. Kariadi General Hospital Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: No.16373/EC/KEPK-RSDK/2025
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Biliary Atresia; Kasai Portoenterostomy; Mesenchymal Stem Cell Transplantation; Liver Function Disorders; Liver Fibrosis; Survival Rate
MeSH Terms: conditions — Biliary Atresia; Liver Cirrhosis | interventions — Portoenterostomy, Hepatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (UC-MSC Group) (Experimental): Participants in this group are infants diagnosed with biliary atresia who undergo Kasai portoenterostomy before 90 days of age. During the operation, they receive intraoperative trans-portal vein injection of umbilical cord-derived mesenchymal stem cells (UC-MSCs) at a dose of 20 million cells diluted in 5 mL autologous plasma.
  Interventions: Biological: Umbilical Cord-Derived Mesenchymal Stem Cells (UC-MSCs); Procedure: Kasai Portoenterostomy
- Control Group (Historical Control Group) (Placebo Comparator): Participants in this group are historical patients who previously underwent Kasai portoenterostomy before 90 days of age at the same institution but did not receive UC-MSC therapy. Data for this group is collected retrospectively.
  Interventions: Procedure: Kasai Portoenterostomy

INTERVENTIONS:
Biological: Umbilical Cord-Derived Mesenchymal Stem Cells (UC-MSCs) — Intraoperative trans-portal vein injection of 20 million mesenchymal stem cells derived from umbilical cord tissue, suspended in 5 mL autologous plasma.
  Arms: Intervention Group (UC-MSC Group)
Procedure: Kasai Portoenterostomy — Surgical procedure to create a portoenterostomy for biliary drainage in infants with biliary atresia.

SUMMARY:
The goal of this clinical trial with historical control is to evaluate whether umbilical cord-derived mesenchymal stem cell (UC-MSC) therapy can improve clinical outcomes in infants with biliary atresia undergoing Kasai surgery before 90 days of age.

The main questions it aims to answer are:

Does UC-MSC therapy improve liver function parameters (bilirubin, albumin, liver enzymes, coagulation profile)? Does UC-MSC therapy reduce complications such as anemia, ascites, jaundice, and improve PELD scores? Does UC-MSC therapy improve overall survival compared to standard Kasai surgery alone? Researchers will compare the group receiving UC-MSC in 2025-2027 with a historical control group of patients who previously underwent Kasai surgery without UC-MSC therapy.

Participants will:

Undergo preoperative evaluation, including laboratory and imaging tests. Receive Kasai surgery combined with intraoperative trans-portal vein injection of 20 million UC-MSCs.

Be monitored postoperatively through serial laboratory tests, imaging (Fibroscan), and clinical assessments at scheduled intervals.

Be followed up for potential serious adverse events and survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Infants diagnosed with biliary atresia confirmed by intraoperative findings.
* Underwent Kasai portoenterostomy at an age less than 90 days.
* Parents or legal guardians have provided informed consent to participate in the study and follow all study procedures.

Exclusion Criteria:

* Infants with severe malnutrition.
* Infants with major congenital anomalies other than biliary atresia.
* Infants with positive tumor markers.

Ages: 0 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2025-06-17 (Estimated); Primary Completion 2026-04-17 (Estimated); Study Completion 2026-04-17 (Estimated)

PRIMARY OUTCOMES:
Serum Albumin Level | Baseline (Pre-op), 4 weeks, 6 weeks, 12 weeks, 24 weeks, and 12 months post-operation
  Measurement of serum albumin as marker of liver synthetic function
Total Bilirubin Level | Baseline, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 12 months
  Measurement of bilirubin levels (total, direct, indirect)
Gamma Glutamyl Transferase (GGT) | Baseline, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 12 months
  Measurement of liver enzyme levels
Alanine Aminotransferase (ALT) | Baseline, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 12 months
  Liver injury marker
Aspartate Aminotransferase (AST) | Baseline, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 12 months
  Liver injury marker
Prothrombin Time (PT), aPTT, INR | Baseline, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 12 months
  Coagulation parameters
Alpha Fetoprotein (AFP) | Baseline, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 12 months
  Tumor marker
Alkaline Phosphatase (ALP) | Baseline, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 12 months
  Liver and bone function marker
Lactate Dehydrogenase (LDH) | Baseline, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 12 months
  Tissue injury marker

SECONDARY OUTCOMES:
Anemia Status | Baseline, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 12 months
  Clinical and laboratory evaluation of anemia
Ascites | Baseline, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 12 months
  Clinical evaluation via physical exam and ultrasound
Jaundice Status | Baseline, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 12 months
  Clinical and laboratory bilirubin assessment
Pediatric End-Stage Liver Disease (PELD) Score | Baseline, 4 weeks, 6 weeks, 12 weeks, 24 weeks, 12 months
  Disease severity scoring system
Overall Survival (OS) | From the surgery date up to the end of the study (12 months maximum follow-up)
  Survival rate since intervention

CONTACTS AND LOCATIONS:
Overall Officials: Avriana Pety Wardani, MD, Sp.BA, Principal Investigator — Dr. Kariadi General Hospital Medical Center; Erik Prabowo, Dr, MD, M.Si.Med, Sp.B-KBD, Study Director — Dr. Kariadi General Hospital Medical Center; Kevin Christian Tjandra, MD, Study Chair — Universitas Diponegoro; Danendra Rakha Putra Respati, MD, Study Chair — Universitas Diponegoro
Locations (1):
- Dr. Kariadi General Hospital Medical Center, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available. The individual participant data will not be shared due to privacy concerns and ethical considerations related to the protection of identifiable health information of pediatric patients. Data sharing is also restricted by institutional policy and local regulations.